CLINICAL TRIAL: NCT04284098
Title: Ultrasound Guided Pectoral Nerve Block Using Bupivacaine Versus Bupivacaine and Dexmedetomidine as a Supplement to General Anesthesia in Modified Radical Mastectomy
Brief Title: PECS Block With Bupivacaine Vs Bupivacaine and Dexmedetomidine in Modified Radical Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Thorya Mohammed Salem, Principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PECS in Breast Cancer Surgery
Record Dates: First submitted 2020-02-14; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Anesthesia, General; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GA group (Placebo Comparator): Group I (GA group): Standard general anesthesia (GA) .
  Interventions: Other: General anesthesia (GA).
- Bupivacaine group (Active Comparator): Group II (B group): ultrasound-guided PECS block using bupivacaine 0.25% + standard GA.
  Interventions: Other: PECS block using bupivacaine .
- Dexmedetomidine&bupivacaine group (Active Comparator): Group III (D group): ultrasound-guided PECS block using bupivacaine 0.25% and Dexmedetomidine 1µg/kg+standard GA.
  Interventions: Other: PECS block using bupivacaine and dexmedetomidine

INTERVENTIONS:
Other: General anesthesia (GA). — Patients received standard GA including fentanyl as intraoperative analgesic and morphine as postoperative analgesic in the first 24 hours.
  Arms: GA group
Other: PECS block using bupivacaine . — The patients undergo an ultrasound-guided PECS I using 10 ml bupivacaine 0.25% and PECS II using 20 ml bupivacaine 0.25%, after 10-minutes observation the patients receive standard GA including fentanyl as intraoperative analgesic and morphine as postoperative analgesic in the first 24 hours.
  Arms: Bupivacaine group
Other: PECS block using bupivacaine and dexmedetomidine — D group:The patients undergo an ultrasound-guided PECS I using 10 ml bupivacaine 0.25% and PECS II using 20 ml bupivacaine 0.25%+dexmedetomidine (1µg/kg) after 10-minutes observation the patients receive standard GA including fentanyl as intraoperative analgesic and morphine as postoperative analgesic in the first 24 hours.
  Arms: Dexmedetomidine&bupivacaine group

SUMMARY:
The incidence of breast cancer as well as the need for surgical treatment has increased.

Breast cancer surgery (BCS) is associated with many complications such as increased incidence of acute and chronic postoperative pain, postoperative nausea and vomiting (PONV), delayed hospital discharge.

Acute postoperative pain is an integral risk factor in the development of chronic pain after BCS.

Inadequate pain control can impact patient recovery including impaired pulmonary and immune function with an increased risk of ileus, thromboembolism, and myocardial infarction.

General anesthesia (GA) is the technique that commonly used for breast surgeries. The downside of GA includes inadequate pain control with high incidence of PONV . Also postoperative opioid for postoperative pain usually associated with many complications Regional anesthesia for breast surgery holds a great promise for breast cancer patients in terms of improved acute pain control with chronic pain prevention. It offers adequate analgesia while minimizing opioid consumption.

This study was designed in order to assess the efficacy and safety of PECS block as a supplement to GA in modified radical mastectomy (MRM) . Also to assess its role in decreasing the amount of opioid in the intra- and postoperative period after MRM. Also to assess its role in decreasing postoperative complications after BCS such as postoperative nausea and vomiting, delayed hospital discharge,and acute postoperative pain. Also to assess the role of dexmedetomidine in prolongation of the analgesic effect of PECS block.

DETAILED DESCRIPTION:
Breast cancer is the most frequent cancer among women; it causes the highest number of cancer-related deaths among them globally. The prognosis has improved considerably over the past 30 years, and the 5-year survival rate of patients has been increased due to the advances in the early detection and treatment of breast cancer.

Breast cancer surgery is associated with many complications such as increased incidence of acute and chronic postoperative pain, postoperative nausea and vomiting, delayed hospital discharge, and cancer recurrence. One of the most important complications is the occurrence of acute postoperative pain. Acute postoperative pain is an integral risk factor in the development of chronic pain after breast cancer surgery (BCS).

Inadequate pain control can impact patient recovery including impaired pulmonary and immune function with an increased risk of ileus, thromboembolism, and myocardial infarction. These factors can further increase the hospital length of stay, increase the healthcare costs, and decrease the patient satisfaction.

General anesthesia, including intravenous and inhalational agents, is the technique that commonly used for breast surgeries. The drawbacks of general anesthesia include inadequate pain control with high incidence of nausea and vomiting. Also the use of opioid and non-opioid analgesics for postoperative pain usually associated with many complications.

Regional anesthesia for breast surgery holds a great promise for breast cancer patients in terms of improved acute pain control with chronic pain prevention. It offers adequate analgesia while minimizing opioid consumption and its related side effects.

Several techniques of blocks for breast surgery have been described. Thoracic epidural and paravertebral blocks were the gold standard techniques to achieve this goal. However, these techniques are generally performed before general anesthesia, and not all anesthesiologists feel comfortable using such invasive procedures in BCS. AS an alternative for these techniques, pectoral nerves (PECS) block has been reported as a promising technique during BCS.

PECS block is an interfascial peripheral nerve block described since 2011.The original block is PECS I block, in which local anesthetic is deposited between the pectoralis major and pectoralis minor muscles to block the lateral pectoral nerve (C5, 6, 7) and medial pectoral nerve (C8, T1) providing analgesia to the anterior chest wall.

PECS II block is a modified PECS I. In this block, local anesthetic is injected between the serratus anterior and pectoralis minor muscle at the third rib in addition to the original block aimed to block thoracic intercostal nerves (T2-6) including intercostobrachial nerve and long thoracic nerve (C5-C7). This modification aimed to extend analgesia to the axilla; this is needed for axillary clearance, necessary for wide excisions, tumorectomy, lymph node excision and several types of mastectomies.

It differs from thoracic epidural and paravertebral blocks as there is no associated sympathetic block. It can be performed while the patient in the supine position and it can be done before or after induction of general anesthesia.

The use of ultrasound (US) makes the pectoral nerve block more accurate and less injurious to nearby structures such as the parietal pleura. It helps direct visualization of anatomical structures, it finds the possible variations in the origin, course, the accompanying structures of the medial and lateral pectoral nerves and their relation to the important structures such thoracoacromial artery and parietal pleura to avoid their injury during performing the PECS block.

The addition of dexmedetomidine to bupivacaine can improve the quality of the block, significantly prolong the duration of analgesia, and provides better pain control postoperatively without major side effects.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized for modified radical mastectomy. American Society of Anesthesiologists (ASA), physical status II. Age between 21-65 year.

Exclusion Criteria:

Patient's refusal. Preexisting coagulopathy or anti-coagulant therapy. Local infection at site of injection. Pregnancy or breast feeding. Body Mass Index (BMI) > 35kg/m². Allergy to local anesthetics and drugs used. Prior breast surgery except for diagnostic biopsies.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Total intraoperative opioid consumption. | During operation.
  Total intraoperative fentanyl.
Total postoperative opioid consumption. | First 24 hours after surgery.
  Total postoperative morphine consumption.
First time to rescue analgesia. | First 24 hours after surgery.
  Duration of postoperative analgesia.

SECONDARY OUTCOMES:
Postoperative pain score. | 0.3,6,9,12, and 24 hours after surgery.
  Visual analogue scale (VAS) which is a unidimensional measure of pain intensity, it is a 10 cm line ranging from (0=no pain to 10 = worst pain imaginable) . The patient is asked to mark on this line where the intensity of the pain lies.
Postoperative nausea &vomiting | First 24 hours after surgery.
  postoperative nausea &vomiting (yes or no)
Hospital length of stay. | First 3 days after surgery.
  days until the patients are discharged to home.
Patients and surgeon satisfaction | First 24 hours after surgery.
  Surgeon satisfaction is assessed by Surgeon Satisfaction with Anesthesia Services (SSAS) the scale was composed of four levels (Strongly disagree, Disagree, Agree, strongly agree) ,Patient satisfaction (yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Doaa M Farid, MD, Study Chair — Faculty of medicine,Zagazig university,Egypt; Maha I El desouky, MD, Study Chair — Faculty of medicine,Zagazig university,Egypt; Fatma M Ahmed, MD, Study Director — Faculty of medicine,Zagazig university,Egypt
Locations (1):
- Thorya M Salem, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battista C, Krishnan S. Pectoralis Nerve Block. 2023 Jul 25. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK547691/ PMID 31613471
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Besch G, Lagrave-Safranez C, Ecarnot F, De Larminat V, Gay C, Berthier F, Samain E, Pili-Floury S. Pectoral nerve block and persistent pain following breast cancer surgery: an observational cohort study. Minerva Anestesiol. 2018 Jun;84(6):769-771. doi: 10.23736/S0375-9393.18.12544-2. Epub 2018 Feb 15. No abstract available. PMID 29469548
- [Background] Campos M, Azevedo J, Mendes L, Rebelo H. Pectoral nerve block as a single anesthetic technique for breast surgery and sentinel lymph node investigation. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Nov;65(9):534-536. doi: 10.1016/j.redar.2018.05.005. Epub 2018 Jul 21. English, Spanish. PMID 30037430
- [Background] Turbitt L, Nelligan K, McCartney C. Pectoral Nerve Blocks for Breast Cancer Surgery: A Methodological Evaluation. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):388-9. doi: 10.1097/AAP.0000000000000226. No abstract available. PMID 26079354